CLINICAL TRIAL: NCT05410444
Title: Application of Intermittent Catheterization in Patients With Micturition Dysfunction After Postoperative Radiotherapy for Cervical Cancer
Brief Title: The Role of Clean Intermittent Catheterization in Patients Undergoing Radiotherapy After Radical Hysterectomy for Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yin ZhuoMin, MD, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZJCH-RCT
Record Dates: First submitted 2022-06-02; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical cancer; Radiotherapy; Clean intermittent catheterization; Bladder function
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Intermittent Urethral Catheterization

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Active Comparator): The control group received routine indwelling catheterization, the catheter was continuously opened, and the indwelling catheter was replaced every 7 days. When the bladder function returned to normal, the catheter was removed.
  Interventions: Device: Indwelling catheterization
- The study group (Experimental): The observation group, namely intermittent catheterization group, was given one-to-one training and education to patients and their families before the implementation of the project. Frequency and timing of intermittent catheterization: it is recommended to catheterize once every 4 hours and no more than 6 times every 24 hours. If the residual urine volume decreases, the number of catheterization can be appropriately reduced; Before each catheterization, urinate by yourself. The derived urine volume is the residual urine volume. The total amount of urine shall not exceed the safe capacity of the bladder.
  Interventions: Device: Clean Intermittent Catheterization

INTERVENTIONS:
Device: Clean Intermittent Catheterization — Under clean conditions, the method of regularly inserting the urinary catheter into the bladder through the urethra and emptying the urine regularly is called clean intermittent catheterization.
  Arms: The study group
Device: Indwelling catheterization — A catheter is inserted into the bladder through the urethra to drain urine. The catheter has been left in the patient's body.
  Arms: The control group

SUMMARY:
Through a prospective, randomized and controlled research design method, this study implemented intermittent catheterization for patients with urinary dysfunction after postoperative radiotherapy of cervical cancer, formulated a reasonable bladder rehabilitation training plan, reduced the amount of residual urine, restored bladder function as soon as possible, reduced the incidence of urinary complications and readmission rate, and improved the quality of life of patients, To comprehensively evaluate the application value of intermittent catheterization in patients with micturition dysfunction after postoperative radiotherapy for cervical cancer.

DETAILED DESCRIPTION:
In this study, patients with postoperative radiotherapy for cervical cancer complicated with voiding dysfunction in the Department of gynecology and oncology radiotherapy of our hospital from July 2018 to December 2020 were selected as the research objects. At the beginning of the study, a total of 80 people were randomly divided into two groups: 40 cases in the observation group and 40 cases in the control group. The observation group implemented intermittent catheterization and formulated a reasonable bladder rehabilitation training plan, and the control group received routine indwelling catheterization. The observation group gave one-to-one training and education to patients and their families before the implementation of the project, including 1. Watching the operation video of intermittent catheterization for female patients. 2. The nurse demonstrated on the simulator. 3. Distribution of drinking water and urination plan, such as paper urination plan, etc. Drinking water plan: patients are required to drink about 1800ml-2000ml of water every day, including drinking water, soup, fruit, etc. it is recommended that the water intake for three meals in the morning, noon and evening is 400ml respectively, and about 200ml water is taken between meals. 200ml water is taken 2 hours after dinner, and no water is taken 2-3 hours before going to bed. Frequency and timing of intermittent catheterization: it is recommended to catheterize once every 4 hours and no more than 6 times every 24 hours. If the residual urine volume decreases, the number of catheterization can be appropriately reduced; Before each catheterization, urinate by yourself. The derived urine volume is the residual urine volume. The total amount of urine shall not exceed the safe capacity of the bladder. 4. The nurse guides the catheterization with hands on the patient until the patient or family members fully master the operation. 5. Nurses add wechat to patients or their families to answer patients' questions and solve operational problems at any time; For three consecutive days after the beginning of intermittent catheterization, patients need to take photos and upload their drinking water and urination diaries every day. Nurses assess the existing risks and deficiencies, give guidance and continue to follow up. 6. If the residual urine volume of the patient is less than 100ml or less than 20% of the safe capacity of the bladder for 3 consecutive days, it is judged that the bladder function has been restored and intermittent catheterization can be stopped. 7. In case of adverse events during the implementation of the project, such as urinary tract infection and impaired renal function, it is necessary to communicate with the doctor in time to decide whether to continue intermittent catheterization. During radiotherapy, the bladder function of the observation group and the control group was evaluated every 7 days until the end of radiotherapy. All patients need to fill in SF-36 questionnaire before and after radiotherapy. In principle, the questionnaire star or paper questionnaire is required to be filled in by the patients themselves. For those who can communicate but can not read and fill in by themselves, the family members shall assist in completing it together. All options of the scale are required to be the opinions of the patients themselves. Drinking water and urination diary records shall be completed by patients and their families. The general information of patients is completed by medical staff at the end of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 and younger than 65; ② Have normal independent judgment ability; ③ According to the staging standard of International Federation of Obstetrics and gynecology (FIGO) in 2009, the preoperative staging was stage Ⅰ A1 -Ⅱ A2; ④ Patients who need postoperative radiotherapy according to the provisions of NCCN clinical practice guide for cervical cancer in 2015; ⑤ Residual urine volume is more than 100ml.

Exclusion Criteria:

① Extensive hysterectomy with bladder repair; ② Urinary tract infection has occurred at the time of admission / transfer; ③ Hydronephrosis; ④ Patients with contraindications to intermittent catheterization; ⑤ Do not agree to participate in this clinical study; ⑥ Patients with communication difficulties. -

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
the recovery rate of bladder function | 3 years
  At the end of radiotherapy, the recovery rate of bladder function in the observation group was higher than that in the control group (P < 0.05)

SECONDARY OUTCOMES:
the incidence of urinary tract infection | 3 years
  During the radiotherapy, the incidence of urinary tract infection in the observation group was significantly less than that in the control group (P = 0).
the bladder volume | 3 years
  At the end of radiotherapy, the bladder volume of the two groups decreased compared with that before radiotherapy. However, there was no significant difference between two groups (P > 0.05).

CONTACTS AND LOCATIONS:
Overall Officials: wang chunlan, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China,, China